CLINICAL TRIAL: NCT01962441
Title: A Phase 3B Randomized, Open-Label, Multi-Center Trial Assessing Sofosbuvir + Ribavirin for 16 or 24 Weeks and Sofosbuvir + Pegylated Interferon + Ribavirin for 12 Weeks in Subjects With Genotype 2 or 3 Chronic HCV Infection.
Brief Title: SOF (Sovaldi®) +RBV for 16 or 24 Weeks and SOF+RBV+Peg-IFN for 12 Weeks in Adults With Genotype 2 or 3 Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0153; 2013-002641-11 (EudraCT Number)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: 7977; GS-7977; PSI-7977; Sofosbuvir (SOF); Pegylated Interferon (Peg-IFN); Ribavirin (RBV)
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SOF+RBV 16 weeks (Experimental): SOF+RBV for 16 weeks
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 weeks (Experimental): SOF+RBV for 24 weeks
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV+Peg-IFN 12 weeks (Experimental): SOF+RBV+Peg-IFN for 12 weeks
  Interventions: Drug: SOF; Drug: RBV; Drug: Peg-IFN
- Retreatment Substudy (Experimental): Participants from the SOF+RBV arms (16 weeks or 24 weeks) who experienced virologic failure on treatment, or during the posttreatment period at or before Posttreatment Week 24 may be eligible to enroll into the Retreatment Substudy to receive SOF+RBV+Peg-IFN for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: Peg-IFN

INTERVENTIONS:
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
Drug: Peg-IFN — 180 µg administered via subcutaneous injection once weekly
  Arms: Retreatment Substudy; SOF+RBV+Peg-IFN 12 weeks

SUMMARY:
This study will assess the efficacy, safety, and tolerability of 16 or 24 weeks of sofosbuvir (Sovaldi®; SOF) + ribavirin (RBV), and 12 weeks of SOF+RBV+ pegylated interferon (Peg-IFN) in treatment-naive and treatment-experienced adults with chronic genotype 3 hepatitis C virus (HCV) infection, and treatment-experienced adults with cirrhosis and chronic genotype 2 HCV infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, age greater than or equal to 18 years.
* Confirmed chronic HCV infection.
* Subjects will have cirrhosis status assessment; liver biopsy may be required.
* Genotype 2 subjects must have cirrhosis of the liver to be eligible.
* Treatment-naive or prior treatment failure to ≥12 weeks of an interferon- based regimen that was not discontinued prematurely due to an adverse event
* Infection with HCV genotype 2 or 3 as determined at Screening
* Body mass index (BMI) greater than or equal to 18 kg/m^2
* Screening laboratory values within predefined thresholds.
* Liver imaging (e.g., ultrasound) within 6 months of Baseline/Day 1 is required in cirrhotic patients to exclude hepatocellular carcinoma (HCC). In the event of intrahepatic lesions, triple phase CT scan or MRI should be performed to exclude HCC.
* Subject must be of generally good health as determined by the Investigator.

Key Exclusion Criteria:

* Prior use of any other inhibitor of the HCV nonstructural protein (NS)5B polymerase
* Pregnant or nursing female or male with pregnant female partner
* History of any other clinically significant chronic liver disease.
* HIV or chronic hepatitis B virus (HBV) infection.
* Malignancy with the exception of certain resolved skin cancers.
* Chronic use of systemically administered immunosuppressive agents.
* Clinically-relevant drug or alcohol abuse.
* History of solid organ transplantation.
* Current or prior history of clinical hepatic decompensation.
* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
* Known hypersensitivity to interferon, RBV, the study investigational medicinal product, the metabolites, or formulation excipients.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (67):
- United States (22):
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Miami, Florida
  - Wellington, Florida
  - Marietta, Georgia
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Novi, Michigan
  - Saint Paul, Minnesota
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Binghamton, New York
  - New York, New York
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Norfolk, Virginia
  - Seattle, Washington
- Australia (12):
  - Camperdown, New South Wales
  - Kogarah, New South Wales
  - Westmead, New South Wales
  - Brisbane, Queensland
  - Greenslopes, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Nedlands Perth, Western Australia
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- New Zealand (4):
  - Grafton, Auckland
  - Christchurch, Chatham Islands
  - Hamilton, Waikato Region
  - Wellington
- United Kingdom (19):
  - Edgbaston, Birmingham
  - Cambridge, Cambridgeshire
  - London, LN
  - Birmingham
  - Bradford
  - Dundee
  - Edinburgh
  - Frimley
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Nottingham
  - Oxford
  - Plymouth
  - Portsmouth
  - Southampton

REFERENCES:
- [Result] Foster GR, Pianko S, Brown A, Forton D, Nahass RG, George J, Barnes E, Brainard DM, Massetto B, Lin M, Han B, McHutchison JG, Subramanian GM, Cooper C, Agarwal K; BOSON Study Group. Efficacy of sofosbuvir plus ribavirin with or without peginterferon-alfa in patients with hepatitis C virus genotype 3 infection and treatment-experienced patients with cirrhosis and hepatitis C virus genotype 2 infection. Gastroenterology. 2015 Nov;149(6):1462-70. doi: 10.1053/j.gastro.2015.07.043. Epub 2015 Aug 4. PMID 26248087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, North America, Australia, and New Zealand. The first participant was screened on 24 September 2013. The last study visit occurred on 07 July 2016.
Pre-assignment Details: 776 participants were screened.
Groups:
- SOF+RBV 16 Weeks, Then Retreatment: Randomized Period: Sofosbuvir (Sovaldi®; SOF) 400 mg tablet administered orally once daily + ribavirin (RBV) tablets administered orally (1000 or 1200 mg daily based on weight) for 16 weeks
  Retreatment Period: Participants who experienced virologic failure during treatment or relapsed at or before Posttreatment Week 24 during the Randomized Period were eligible to enroll into the Retreatment Period to receive SOF+Peg-IFN+RBV for 12 weeks.
- SOF+RBV 24 Weeks, Then Retreatment: Randomized Period: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 24 weeks
  Retreatment Period: Participants who experienced virologic failure during treatment or relapsed at or before Posttreatment Week 24 during the Randomized Period were eligible to enroll into the Retreatment Period to receive SOF+Peg-IFN+RBV for 12 weeks.
- SOF+RBV+Peg-IFN 12 Weeks: Randomized Period: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) + pegylated interferon (Peg-IFN) 180 µg administered subcutaneously once weekly for 12 weeks
  Participants in this group were not eligible to enroll into the Retreatment Period.
Period: Randomized Period
Arm/Group | SOF+RBV 16 Weeks, Then Retreatment | SOF+RBV 24 Weeks, Then Retreatment | SOF+RBV+Peg-IFN 12 Weeks
Started | 200 | 201 | 200
Completed | 190 | 190 | 189
Not Completed | 10 | 11 | 11
Not completed — Randomized but Never Treated | 4 | 2 | 3
Not completed — Lost to Follow-up | 2 | 4 | 4
Not completed — Withdrew Consent | 3 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Period: Retreatment Substudy
Arm/Group | SOF+RBV 16 Weeks, Then Retreatment | SOF+RBV 24 Weeks, Then Retreatment | SOF+RBV+Peg-IFN 12 Weeks
Started | 20 (20 participants who experienced virologic failure enrolled into the Retreatment Substudy.) | 10 (10 participants who experienced virologic failure enrolled into the Retreatment Substudy.) | 0 (Participants in the SOF+RBV+Peg-IFN group were not eligible to enroll in the Retreatment Substudy.)
Completed | 18 | 10 | 0
Not Completed | 2 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants with genotype 2 or 3 HCV infection who were randomized and received at least 1 dose of study drug.
Groups:
- SOF+RBV 16 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 16 weeks
- SOF+RBV 24 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 24 weeks
- SOF+RBV+Peg-IFN 12 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) + Peg-IFN 180 µg administered subcutaneously once weekly for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks | Total
Number analyzed (Participants) | 196 | 199 | 197 | 592
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.7) | 49 (9.8) | 50 (10.2) | 50 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 70 | 65 | 197
  Male | 134 | 129 | 132 | 395
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 5 | 2 | 12
  Not Hispanic or Latino | 188 | 188 | 191 | 567
  Not Disclosed | 3 | 6 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2 | 2 | 2 | 6
  White | 162 | 168 | 165 | 495
  Asian | 29 | 26 | 25 | 80
  American Indian/ Alaska Native/ First Nations | 2 | 0 | 0 | 2
  Hawaiian or Pacific Islander | 0 | 1 | 2 | 3
  Other | 0 | 1 | 1 | 2
  Not Disclosed | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  New Zealand | 15 | 12 | 13 | 40
  Canada | 21 | 33 | 29 | 83
  United States | 29 | 33 | 31 | 93
  United Kingdom | 86 | 82 | 80 | 248
  Australia | 45 | 39 | 44 | 128
HCV Genotype [Number; unit: participants]
  Genotype 2 | 15 | 17 | 16 | 48
  Genotype 3 | 181 | 182 | 181 | 544
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 75 | 73 | 78 | 226
    CT | 94 | 95 | 98 | 287
    TT | 27 | 31 | 21 | 79
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.68) | 6.2 (0.71) | 6.3 (0.69) | 6.3 (0.69)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 60 | 72 | 60 | 192
  ≥ 6 log10 IU/mL | 136 | 127 | 137 | 400

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 196 | 199 | 197
percentage of participants | 71.9 | 85.4 | 92.9

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 196 | 199 | 197
percentage of participants | 1.5 | 1.5 | 1.5

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 196 | 199 | 197
percentage of participants
  SVR4 | 73.0 | 85.9 | 95.9
  SVR24 | 71.9 | 84.4 | 93.4

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 196 | 199 | 197
percentage of participants
  Week 1 | 14.8 | 20.1 | 25.9
  Week 2: number analyzed (Participants) | 195 | 198 | 197
  Week 2 | 53.3 | 53.5 | 67.0
  Week 4: number analyzed (Participants) | 194 | 198 | 195
  Week 4 | 86.6 | 91.9 | 97.4
  Week 8: number analyzed (Participants) | 193 | 198 | 195
  Week 8 | 99.5 | 99.5 | 99.5
  Week 12: number analyzed (Participants) | 190 | 197 | 194
  Week 12 | 100.0 | 98.5 | 100.0
  Week 16: number analyzed (Participants) | 191 | 194 | 0
  Week 16 | 99.0 | 99.5 |
  Week 20: number analyzed (Participants) | 0 | 194 | 0
  Week 20 |  | 99.5 |
  Week 24: number analyzed (Participants) | 0 | 193 | 0
  Week 24 |  | 100.0 |

5. Secondary Outcome: HCV RNA at Weeks 1, 2, 4, 8, and 12
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 194 | 198 | 195
log10 IU/mL
  Week 1: number analyzed (Participants) | 194 | 197 | 194
  Week 1 | 2.13 (0.658) | 2.08 (0.749) | 1.81 (0.576)
  Week 2: number analyzed (Participants) | 191 | 196 | 195
  Week 2 | 1.44 (0.436) | 1.45 (0.487) | 1.32 (0.342)
  Week 4: number analyzed (Participants) | 193 | 198 | 195
  Week 4 | 1.19 (0.156) | 1.21 (0.287) | 1.16 (0.085)
  Week 8: number analyzed (Participants) | 193 | 198 | 194
  Week 8 | 1.15 (0.021) | 1.15 (0.100) | 1.15 (0.000)
  Week 12: number analyzed (Participants) | 191 | 197 | 194
  Week 12 | 1.15 (0.000) | 1.17 (0.318) | 1.15 (0.000)

6. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 8, and 12
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 194 | 198 | 195
log10 IU/mL
  Week 1: number analyzed (Participants) | 194 | 197 | 194
  Week 1 | -4.18 (0.559) | -4.15 (0.664) | -4.46 (0.556)
  Week 2: number analyzed (Participants) | 191 | 196 | 195
  Week 2 | -4.86 (0.661) | -4.78 (0.714) | -4.96 (0.661)
  Week 4: number analyzed (Participants) | 193 | 198 | 195
  Week 4 | -5.11 (0.671) | -5.02 (0.735) | -5.12 (0.699)
  Week 8: number analyzed (Participants) | 193 | 198 | 194
  Week 8 | -5.16 (0.684) | -5.08 (0.708) | -5.12 (0.691)
  Week 12: number analyzed (Participants) | 191 | 197 | 194
  Week 12 | -5.15 (0.686) | -5.05 (0.788) | -5.12 (0.691)

7. Secondary Outcome: Percentage of Participants Experiencing On-Treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 196 | 199 | 197
percentage of participants | 0 | 1.5 | 0

8. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse is defined as HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 195 | 195 | 195
percentage of participants | 26.7 | 12.3 | 4.6

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days (Randomized Period) Up to 12 additional weeks plus 30 days (Retreatment Period)
Description: Safety Analysis Set: participants with genotype 2 or 3 HCV infection who were randomized and received at least 1 dose of study drug.
  MedDRA version 18.0 = Randomized Period; MedDRA version 19.0 = Retreatment Period
Groups:
- Randomized Period: SOF+RBV 16 Weeks: Randomized Period: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 16 weeks
- Randomized Period: SOF+RBV 24 Weeks: Randomized Period: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 24 weeks
- Randomized Period: SOF+RBV+Peg-IFN 12 Weeks: Randomized Period: SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) + Peg-IFN 180 µg administered subcutaneously once weekly for 12 weeks
- Retreatment Period: SOF+RBV+Peg-IFN 12 Weeks: Retreatment Period: Participants from the SOF+RBV 16 Weeks or 24 Weeks groups who experienced virologic failure during treatment or relapsed at or before Posttreatment Week 24 during the Randomized Period were eligible to enroll into the Retreatment Period to receive SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) + Peg-IFN 180 µg administered subcutaneously once weekly for 12 weeks.
Arm/Group | Randomized Period: SOF+RBV 16 Weeks | Randomized Period: SOF+RBV 24 Weeks | Randomized Period: SOF+RBV+Peg-IFN 12 Weeks | Retreatment Period: SOF+RBV+Peg-IFN 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/199 | 0/197 | 0/30
Serious Adverse Events (participants affected / at risk) | 8/196 | 10/199 | 12/197 | 1/30
Other Adverse Events (participants affected / at risk) | 173/196 | 176/199 | 192/197 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Period: SOF+RBV 16 Weeks (N=196) | Randomized Period: SOF+RBV 24 Weeks (N=199) | Randomized Period: SOF+RBV+Peg-IFN 12 Weeks (N=197) | Retreatment Period: SOF+RBV+Peg-IFN 12 Weeks (N=30)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Miscarriage of partner (Social circumstances) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Period: SOF+RBV 16 Weeks (N=196) | Randomized Period: SOF+RBV 24 Weeks (N=199) | Randomized Period: SOF+RBV+Peg-IFN 12 Weeks (N=197) | Retreatment Period: SOF+RBV+Peg-IFN 12 Weeks (N=30)
Anaemia (Blood and lymphatic system disorders) | 4 | 7 | 12 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 11 | 2
Dry eye (Eye disorders) | 3 | 5 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 8 | 11 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 10 | 9 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 18 | 27 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 7 | 12 | 0
Dyspepsia (Gastrointestinal disorders) | 10 | 12 | 11 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 8 | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 5 | 3 | 5 | 2
Nausea (Gastrointestinal disorders) | 32 | 34 | 50 | 7
Vomiting (Gastrointestinal disorders) | 10 | 21 | 19 | 0
Asthenia (General disorders) | 2 | 3 | 10 | 0
Chills (General disorders) | 3 | 4 | 21 | 1
Fatigue (General disorders) | 74 | 83 | 92 | 18
Influenza like illness (General disorders) | 7 | 8 | 39 | 6
Injection site rash (General disorders) | 0 | 0 | 5 | 2
Pyrexia (General disorders) | 5 | 7 | 29 | 6
Nasopharyngitis (Infections and infestations) | 12 | 14 | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 10 | 3 | 0
Platelet count decreased (Investigations) | 0 | 0 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 13 | 16 | 35 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15 | 25 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 14 | 15 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 22 | 11 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 19 | 33 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 11 | 16 | 13 | 2
Dizziness postural (Nervous system disorders) | 3 | 1 | 10 | 0
Dysgeusia (Nervous system disorders) | 6 | 4 | 10 | 1
Headache (Nervous system disorders) | 61 | 72 | 70 | 12
Lethargy (Nervous system disorders) | 9 | 8 | 10 | 1
Memory impairment (Nervous system disorders) | 10 | 3 | 5 | 1
Anxiety (Psychiatric disorders) | 12 | 16 | 17 | 1
Depressed mood (Psychiatric disorders) | 8 | 11 | 17 | 0
Depression (Psychiatric disorders) | 1 | 8 | 10 | 3
Insomnia (Psychiatric disorders) | 47 | 56 | 50 | 2
Irritability (Psychiatric disorders) | 17 | 25 | 21 | 3
Mood swings (Psychiatric disorders) | 3 | 7 | 5 | 3
Sleep disorder (Psychiatric disorders) | 15 | 7 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 19 | 28 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 22 | 22 | 30 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 12 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 9 | 16 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 22 | 25 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 24 | 22 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 9 | 16 | 15 | 0
Rash (Skin and subcutaneous tissue disorders) | 24 | 27 | 39 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years